CLINICAL TRIAL: NCT03052231
Title: Evaluating the Feasibility of Interactive Mobile Health Information to Enhance Patient Care at a Cystic Fibrosis Center
Brief Title: Interactive Mobile Health Information to Enhance Patient Care at a Cystic Fibrosis Center
Acronym: MOMMI3CFCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landon Pediatric Foundation (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LandonPF
Record Dates: First submitted 2015-12-24; First posted 2017-02-14 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Medication Adherence; Cystic Fibrosis
Keywords: adherence; cystic fibrosis
MeSH Terms: conditions — Medication Adherence; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interactive Mobile Health Information (Active Comparator): Receives Interactive Mobile Health Information via caremessage. EAI staff focus group content will include qualitative descriptions of their experiences with training and actual use of the Caremessages.org service, as well as to elicit comments about contributing features and other mitigating or enhancing factors of the intervention's implementation, outreach and promotion, and integration into workflow practices.
  Interventions: Device: caremessage
- Usual care (No Intervention): Usual care - clinic education, medication refills without reminders, appointments without reminders

INTERVENTIONS:
Device: caremessage — Central to the mobile health information service is the interactive and personalized text-based message system that delivers actionable and tailored health content to participants: office visit appointment reminders; medication adherence reminders; and general health education messages.
  Arms: Interactive Mobile Health Information

SUMMARY:
Real-world adherence to inhaled and oral therapies for cystic fibrosis (CF) patients remains discouragingly low, ranging between 31-53% for inhaled antibiotics and 41-72% for hypertonic saline. Programs to enhance adherence, including comprehensive behavioral interventions with adolescents, have met with mixed success. Advances in therapy, treatment delivery systems, and data capture technology offer the potential for enhancing adherence by providing immediate and more frequent feedback to the patient regarding his or her fidelity to the prescribed treatment regimen. The investigators propose to evaluate a systematic yet technically simple approach to linking treatment and feedback components to enhance adherence in a real-work CF clinic setting that treats a significant minority patient population.

This is the first trial assessing the impact of a collaborative active intervention program of a multi disciplinary team in improving adherence to specific chronic medications and improving clinical outcomes in CF patients. The PI has implemented the texting service (Caremessage.org) with COPD and diabetes patients. The content will be modified to provide both English and Spanish language content relevant to these participants and their standard treatment protocols.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of an interactive mobile health information service in supporting clinic staff (i.e., nurse practitioners, case managers and care coordinators) at a Cystic Fibrosis Center clinic to connect with patients and create conversations around behavior-centered goals. The interactive mobile health information service has been designed to supplement the standard of care by supporting patient-empowerment strategies through:

* educating participants,
* encouraging behavior change, and
* promoting adherence with their treatment protocols.

The project will adapt the iCAN program content as an educational tool to be incorporated in the educational material. iCAN is an electronic platform aimed to provide an engaging environment for diabetic outpatients to self-manage, gain control over their health, and ultimately adhere to their medical appointments and regimen. Similar to diabetes, CF is an all-encompassing chronic disease that requires coordinated efforts among patients, caregivers, and health-care providers across treatment adherence, nutrition, lifestyle choices, and social support systems. Central to the mobile health information service is the interactive and personalized text-based message system that delivers actionable and tailored health content to participants: office visit appointment reminders; medication adherence reminders; and general health education messages. While a number of technically sophisticated applications exist, our approach will involve a less sophisticated and complex approach. Our primary objective is to get the information to the patients, some of whom are members of lower income minority communities. If "simple" interventions prove effective, then the groundwork will have been laid for considering more tailored albeit complex systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Cystic fibrosis at all ages;
* Their associated CF Center professionals;
* Their associated family;
* CF patients that should be treated with one or more of these chronic medications: Tobi (Tobramycin), (Colistin), Pulmozyme (Dornase Alpha), Hypertonic Saline (HS), Creon (pancreatic enzymes), AquaADEKs (Multivitamin);
* Patients willing to participate in a trial;
* Presence of a parent/guardian capable of providing informed consent; and
* Patients attending CF clinic at least once every 12 months.

Exclusion Criteria:

* Absence of a parent/guardian or unwillingness to provide permission;
* Potential participant declines to provide assent; and
* Transplant patients.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of Scheduled appointments attended | Six months
  Secondary objectives include evaluating program processes that enhance participant use of the system: 1) to receive responses to specific questions; 2) to track their individual progress towards achieving health goals, and; 3) to respond to system prompts to self-report data in the interactive component related to their actions or behaviors, e.g. RSVP to appointment reminders, self-management behaviors related to medication adherence, and self-management behaviors related to the achieving health goals. Processes involving program management and impact on barriers to treatment delivery by clinic staff, treating physicians and parents will also be evaluated.

SECONDARY OUTCOMES:
Knowledge of disease Questionnaire | Six Months
  Secondary objectives include evaluating program processes that enhance participant use of the system: 1) to receive responses to specific questions; 2) to track their individual progress towards achieving health goals, and; 3) to respond to system prompts to self-report data in the interactive component related to their actions or behaviors, e.g. RSVP to appointment reminders, self-management behaviors related to medication adherence, and self-management behaviors related to the achieving health goals. Processes involving program management and impact on barriers to treatment delivery by clinic staff, treating physicians and parents will also be evaluated.
FEV1 in LPM | 6 months
  Measure of pulmonary function
Body mass index | six months
  kg/meters squared

CONTACTS AND LOCATIONS:
Overall Officials: Chris Landon, MD, Principal Investigator — Landon Pediatric Foundation
Locations (1):
- Pediatric Diagnostic Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
Share with iCAN

REFERENCES:
- [Background] Eakin MN, Bilderback A, Boyle MP, Mogayzel PJ, Riekert KA. Longitudinal association between medication adherence and lung health in people with cystic fibrosis. J Cyst Fibros. 2011 Jul;10(4):258-64. doi: 10.1016/j.jcf.2011.03.005. Epub 2011 Mar 31. PMID 21458391
- [Background] Quittner A et al. Chest 2011 (4_MeetingAbstracts):908A
- [Background] Imperial College of London. iCAN Self---Management Technology: Helping Patients to Medical Appointments. CID 00884448, May 5, 2014
- [Background] Modi AC, Lim CS, Yu N, Geller D, Wagner MH, Quittner AL. A multi-method assessment of treatment adherence for children with cystic fibrosis. J Cyst Fibros. 2006 Aug;5(3):177-85. doi: 10.1016/j.jcf.2006.03.002. Epub 2006 May 5. PMID 16679071
- [Background] Taddeo D, Egedy M, Frappier JY. Adherence to treatment in adolescents. Paediatr Child Health. 2008 Jan;13(1):19-24. doi: 10.1093/pch/13.1.19. PMID 19119348
- [Background] QSR International, Victoria, Australia, 2015